

# Post-Market Evaluation of the Rotation Medical Rotator Cuff System

**Protocol Number 2014.05.12** 

**REVISION C** 

January 2018

Rotation Medical, Inc.

15350 25th Avenue North Plymouth MN 55447

This study will be conducted in accordance with the protocol and applicable regulatory requirements.

#### **CONFIDENTIAL INFORMATION**

No use or disclosure of information contained within this document is permitted without prior written authorization from Rotation Medical, Inc.

# STUDY CONTACT INFORMATION

# **Study Sponsor:**

Rotation Medical, Inc. 15350 25<sup>th</sup> Avenue North Plymouth, MN 55447

# **Study Contact:**

Jeff Grebner Rotation Medical, Inc. 15350 25<sup>th</sup> Avenue North Plymouth, MN 55447 Phone: (763) 746-7502

Fax: (763) 746-7501

E-mail: jgrebner@rotationmedical.com

# ROTATION MEDICAL, INC. PROTOCOL SIGNATURE PAGE

# Post-Market Evaluation of the Rotation Medical Rotator Cuff System

PROTOCOL NO. 2014.05.12

Revision C

January 2018

I have read this study protocol and the signature below constitutes approval of this protocol and any attachments, and provides the necessary assurances that this study will be conducted in accordance to all stipulations of the protocol and in compliance with applicable local legal and regulatory requirements and applicable U.S. federal regulations including 21 CFR Part 50 (Protection of Human Subjects) and 21 CFR Part 56 (Institutional Review Boards).

| Clinical Site Name | |
|------------------------------------------|------|
| Site Principal Investigator Signature | Date |
| Site Principal Investigator Printed Name | _ |

| PROTOCOL STUDY SYNOPSIS | |
|---|---|
| Title: | Post-Market Evaluation of the Rotation Medical Rotator Cuff System |
| <b>Study Devices:</b> | Rotation Medical Rotator Cuff System <sup>TM</sup> (Cleared for commercial use by the U.S. Food and Drug Administration: K140300; K131637; K131635; K122048) |
| <b>Study Design:</b> | Prospective, non-randomized, post-market study |
| <b>Enrollment:</b> | Up to 150 subjects will be treated |
| Inclusion | |
| Criteria: | <ol> <li>At least 21 years of age</li> <li>Rotator cuff tear requiring surgery that meets either criterion A or B: <ul> <li>A. Medium or large partial-thickness tear or very small full-thickness tear of the supraspinatus tendon planned for standalone treatment (no surgical repair with sutures/suture anchors) with the bioinductive implant</li> <li>B. Medium or large full-thickness tear primarily of the supraspinatus tendon planned for treatment with the bioinductive implant adjunctive to surgical repair</li> </ul> </li> <li>Chronic shoulder pain lasting longer than 3 months unresponsive to conservative therapy including, but not limited to, pain medication, physical therapy and injections</li> <li>MRI of the shoulder within 60 days prior to the study procedure</li> <li>Willing to comply with the prescribed post-operative rehabilitation program</li> <li>Willing to be available for each protocol-required follow-up examination</li> <li>Able to understand the informed consent process, including regulatory requirements such as HIPAA authorization, and document informed consent prior to completion of any study-related procedures</li> <li>Ability to read, understand, and complete subject-reported outcomes in</li> </ol> |
| Exclusion<br>Criteria: | <ol> <li>English</li> <li>Massive rotator cuff tears (≥ 5 cm)</li> <li>Acute rotator cuff tears less than 12 months from injury</li> <li>Previous rotator cuff surgery on the index shoulder</li> <li>Instability of the index shoulder</li> <li>Chondromalacia of index shoulder ≥ Grade 3</li> <li>Fatty infiltration of the index shoulder rotator cuff muscle ≥ Grade 2</li> <li>Calcification of the index shoulder rotator cuff</li> <li>Genetic collagen disease</li> <li>History of insulin dependent diabetes</li> <li>History of auto-immune or immunodeficiency disorders</li> <li>History of chronic inflammatory disorders</li> <li>Oral steroid use in last 2 months or injectable steroid use in last 4 weeks</li> <li>History of heavy smoking (&gt; 1 pack per day) within last 6 months</li> <li>Hypersensitivity to bovine-derived materials</li> <li>Females of child-bearing potential who are pregnant or plan to become pregnant during the course of the study</li> <li>Currently involved in any injury litigation or worker's compensation claims relating to the index shoulder</li> </ol> |

| | 17. Enrolled, or plans to enroll, in another clinical trial during this study that |
|---|---|
| | would affect the outcomes of this study |
| | 18. History of non-compliance with medical treatment, physical |
| | therapy/rehabilitation, or clinical study participation |
| | 19. History of cognitive or mental health status that interferes with study |
| | participation |
| Study | To evaluate bioinduction of new tissue and tendon healing after implantation of |
| <b>Objective:</b> | the Rotation Medical Bioinductive Implant used as either a standalone device or |
| | adjunct to surgical repair in the treatment of supraspinatus tendon tears. |
| Primary | MRI assessment of the following: |
| <b>Outcomes:</b> | 1. Increase in tendon thickness |
| | 2. Integration of induced tissue with the underlying tendon and maturation of |
| | the induced tissue |
| | 3. Amount of defect fill-in and characteristics of both the filled-in tissue within |
| | the tendon tear and underlying tendon (nonsurgically-repaired tears only) |
| | 4. Rotator cuff re-tear rate |
| Secondary | 1. Safety |
| Outcomes: | 2. Procedure parameters |
| | 3. Change in American Shoulder and Elbow Society (ASES) scale |
| | 4. Change in Constant-Murley Shoulder score |
| | 5. Recovery |
| | 6. Subject satisfaction |
| Study | Baseline |
| Assessments | Procedure |
| | Post-procedure follow-up: 3 months, 1 year, 2 years |
| Sponsor: | Rotation Medical, Inc. |
| | 15350 25th Avenue North |
| | Plymouth MN 55447 |
| Data | Rotation Medical, Inc. |
| Management | 15350 25th Avenue North |
| and | Plymouth MN 55447 |
| Monitoring: | 1 Tyllioudi 1viiv 3377/ |

# **TABLE OF CONTENTS**

| 1 | INT | TRODUCTION & RATIONALE | 8 |
|---|---|---|---|
| 2 | DE | EVICE DESCRIPTION | 9 |
| | 2.1 | DEVICE DESCRIPTION | 9 |
| | 2.2 | PRINCIPLES OF OPERATION | 10 |
| 3 | ST | TUDY OBJECTIVE | 10 |
| 4 | ST | UDY DESIGN | 11 |
| | 4.1 | Sample Size | 11 |
| | 4.2 | STUDY DURATION | |
| | 4.3 | PRIMARY OUTCOME MEASURES | |
| | 4.3. | | |
| | 4.3. | 3.2 Integration and Maturation of New Tissue | 11 |
| | 4.3. | | |
| | 4.3. | | |
| | 4.4 | | |
| | 4.4. | | |
| | 4.4.<br>4.4. | | |
| | 4.4.<br>4.4. | | 12 |
| | 4.4.<br>4.4. | | |
| | 4.4. | | |
| 5 | | ATISTICAL ANALYSIS PLAN | |
| J | | Hypothesis Testing, Sample Size and Power | |
| | 5.1<br>5.2 | HYPOTHESIS 1 ESTING, SAMPLE SIZE AND POWER INTERIM ANALYSES | |
| 6 | - | LIGIBILITY CRITERIA | |
| 0 | | | |
| | 6.1 | INCLUSION CRITERIA | |
| | 6.2 | EXCLUSION CRITERIA | |
| 7 | ST | TUDY ASSESSEMENTS | 15 |
| T | ABLE | E 7-1: SCHEDULE OF STUDY ASSESSMENTS | 16 |
| | 7.1 | ELIGIBILITY ASSESSMENT | 16 |
| | 7.2 | ENROLLMENT | 16 |
| | 7.3 | BASELINE ASSESSMENT | |
| | 7.4 | PROCEDURE ASSESSMENT | |
| | 7.5 | PROCEDURE RULES | |
| | 7.6 | POST-OPERATIVE CARE | |
| T | ABLE | E 7-2: POST-OPERATIVE REHABILITATION GUIDELINES | 18 |
| | 7.7 | FOLLOW-UP ASSESSMENTS | |
| | 7.7. | | |
| | 7.7. | | |
| | 7.7. | 1 | |
| | 7.8 | UNSCHEDULED FOLLOW-UP | |
| | 7.9 | REVISION/ADDITIONAL SHOULDER SURGERY | |
| | 7.10<br>7.11 | EARLY WITHDRAWAL OR LOST TO FOLLOW-UP | |
| o | | | |
| 8 | | OVERSE EVENT DEFINITIONS AND REPORTING | |
| | 8.1 | DEFINITION OF ADVERSE EVENT (AE) | 21 |

| 8.2 | SERIOUS ADVERSE EVENT (SAE) | 21 |
|-------|---------------------------------------------------------|----|
| 8.3 | UNANTICIPATED ADVERSE DEVICE EFFECT (UADE) | 22 |
| 8.4 | ASSESSING, RECORDING AND REPORTING AES, SAES, AND UADES | 22 |
| 9 M | IALFUNCTIONS | 22 |
| 10 | PROTOCOL DEVIATIONS | 22 |
| 11 | REPORTING REQUIREMENTS | 23 |
| 12 | RISKS AND BENEFITS | 23 |
| 12.1 | | |
| 12.2 | Benefits | 24 |
| 13 | DATA MANAGEMENT | 24 |
| 13.1 | DATA COLLECTION | 24 |
| 13.2 | DATA PROCESSING | 24 |
| 14 | ADMINISTRATIVE RESPONSIBILITIES | 25 |
| 14.1 | SITE AND INVESTIGATOR SELECTION | 25 |
| 14.2 | | |
| 14.3 | | |
| 14.4 | | |
| 14.5 | | |
| 14.6 | | |
| 14.7 | | |
| 14.8 | | |
| 14.9 | SPONSOR RESPONSIBILITIES | 27 |
| 14.10 | 0 Investigator Responsibilities | 27 |
| 15 | MONITORING AND AUDITING | 28 |
| 16 | REPORTS AND RECORDS | 28 |
| 16.1 | Reports | 28 |
| 16.2 | | |
| 17 | USE OF INFORMATION AND PUBLICATION | 28 |
| 18 | REFERENCES | 28 |

# 1 INTRODUCTION & RATIONALE

Musculoskeletal disorders are one of the most common causes of disability in the United States with approximately 50% of the adult population having experienced a chronic musculoskeletal condition lasting longer than 3 months.<sup>1</sup> After knee-related disorders, shoulders are the second most common joint causing chronic pain with an estimated 18.9 million adults affected. The direct cost of treating shoulder pain is approximately \$7 billion annually and this figure excludes the indirect cost burden (i.e., missed work, lost productivity).<sup>1</sup> With age, the prevalence of rotator cuff disease increases with an estimated 50% of individuals over 66 years of age having bilateral rotator cuff tears.<sup>2,3</sup> Recent demographic and morphological studies of rotator cuff tears also show that these defects increase in size with time and painful tears tend to be larger than asymptomatic tears.<sup>2,4</sup>

Persistent shoulder pain concomitant with a rotator cuff tendon tear is currently treated with arthroscopic subacromial decompression (ASD) with or without cuff repair depending on the size and morphology of the cuff tear. Decompression alone leaves the tendon tear structurally unmodified and does not prevent rotator cuff tear progression. <sup>5,6,7</sup> Cuff repair as a treatment for rotator cuff tears often requires the resection of tendon from the bone and re-attachment using suture anchors. <sup>8,9,10</sup> Estimates of re-tear rates following the completion and repair of small tears have been reported between 10% and 36%. <sup>8,9,11</sup> Peri-operative morbidity and post-operative rehabilitation associated with rotator cuff tendon repair is more extensive for the patient than ASD alone. <sup>7</sup>

The Rotation Medical Bioinductive Implant is a bioabsorbable device that provides a layer of collagen over injured tendons. This device is indicated for the management and protection of tendon injuries in which there has been no substantial loss of tendon tissue and can be implanted either during mini-open or arthroscopic procedures. The device was first evaluated in a preclinical study of 23 sheep that was approved by the Colorado State University Institutional Animal Care and Use Committee. The device did not elicit an inflammatory response or a foreign body reaction and histological analyses confirmed the device was completely absorbed after six months with integration of the new tendinous tissue to the underlying host tendon and a fibrocartilagenous transition zone at the tendon-to-bone insertion site. Tendon thickness at the implant site increased by approximately 2.5 millimeters due to induction of new tendinous tissue and remained stable one year after surgery. <sup>12</sup>

The Rotation Medical Bioinductive Implant was further evaluated in a clinical study of 24 subjects who underwent implantation of the device and completed a minimum of one year follow-up. This study was approved by the Northern Sydney Central Coast Ethics Committee and registered in the Australian New Zealand Clinical Trials Registry [#ACTRN12611001082998]. The procedure was performed arthroscopically in 14 subjects while the other 10 subjects underwent a mini-open procedure. The median implant time was 15 minutes and all subjects were successfully implanted with no intent-to-treat failures. One patient experienced a return to pain 12 months after surgery that was associated with significant bursitis and an arthroscopic clean-up procedure was performed to debride the bursa. Despite the bursal reaction in this patient, tendon healing and tissue induction were not compromised.

Magnetic resonance imaging (MRI) at 3, 6, and 12 months after surgery provided evidence that the device consistently induced the formation of new, tendinous tissue that appeared well-integrated with each patient's native tendon tissue and showed progressive maturation over time. MRI observations were consistent with the histological results from prior sheep studies. <sup>13</sup> Shoulder function and pain was also assessed at 3, 6 and 12 months after treatment using the ASES (American Shoulder and Elbow Surgery) and Constant (Constant-Murley) standard shoulder surveys. <sup>14,15</sup> All of the scores at 12 months were significantly improved from baseline (p < 0.05) and improvement was comparable to published literature. <sup>16</sup>

# 2 DEVICE DESCRIPTION

# 2.1 DEVICE DESCRIPTION

There are three implantable components in the Rotation Medical Rotator Cuff System<sup>TM</sup> (**Figure 2-1**).

- 1. <u>Bioinductive implant:</u> The device is made from highly purified reconstituted collagen fibers derived from bovine tendon and manufactured for Rotation Medical, Inc. by Collagen Matrix, Inc. (Oakland, New Jersey, USA). It is contraindicated for use in patients with a history of hypersensitivity to bovine-derived materials and this is an exclusion criterion for study participation. The device is designed to completely absorb within six to 12 months.
- 2. <u>Tendon staples</u>: The tendon staples are made from poly(L-lactide-co-D,L-lactide) in a molar ratio of 70% L-lactide to 30% D,L-lactide. Polylactide materials have been used in a variety of medical devices, such as bone anchors, bone pins, screws, plates, and spinal fusion cages. The tendon staples are designed to completely absorb within approximately 12 months.
- 3. <u>Bone staples</u>: The bone staples are made from polyetheretherketone (PEEK), which is a common polymer used for bone anchors in orthopedic surgery. The bone staples are not bioabsorbable.

The Rotation Medical Rotator Cuff System has been cleared by the U.S. Food and Drug Administration (FDA) [K140300; K122048; K131635; K131637]. The purpose of this post-market study is to collect and analyze outcomes data under a common protocol.

Bioinductive implant

Bone staple

Tendon staple

Figure 2-1: Rotation Medical Implantable System Components

The tendon and bone staplers used to affix the bioinductive implant to tendon tissue and the head of the humerus respectively are shown in **Figure 2-2**. These are designed as single-use devices.

Figure 2-2: Rotation Medical Single-Use Disposable Staplers



# 2.2 PRINCIPLES OF OPERATION

No investigational devices or procedures will be used in this post-market study and all devices will be used according to their indications for use. Operation, indication, and instructions for use are described in the Instructions for Use (IFUs).

# 3 STUDY OBJECTIVE

To evaluate bioinduction of new tissue and tendon healing after implantation of the Rotation Medical Bioinductive Implant used as either a standalone device or adjunct to surgical repair in the treatment of supraspinatus tendon tears.

# 4 STUDY DESIGN

This is a prospective, non-randomized, single-arm multi-center study conducted under a common protocol designed to evaluate long-term outcomes following arthroscopic or mini-open implantation of the Rotation Medical Bioinductive Implant to treat high-grade partial thickness or small/medium/large (i.e. non-massive) full-thickness rotator cuff tears primarily involving the supraspinatus tendon.

# 4.1 SAMPLE SIZE

Up to 150 subjects will be enrolled and treated with the Rotation Medical Rotator Cuff System at up to 15 study sites in the United States.

# 4.2 STUDY DURATION

Enrollment is anticipated to take up to 12 months and all subjects will be followed for two years after surgery. Therefore, the overall study duration is estimated to be 36 months.

#### 4.3 Primary Outcome Measures

#### 4.3.1 Increase in Tendon Thickness

Supraspinatus tendon thickness will be measured pre-operatively (baseline) and the total thickness of the tendon and any newly induced tissue at the implant site will be measured at each follow-up visit using magnetic resonance imaging (MRI). The mean ( $\pm$  SD) change in post-operative supraspinatus tendon thickness will be calculated at each follow-up interval.

# 4.3.2 Integration and Maturation of New Tissue

Integration and maturation of the newly induced tissue will be assessed by MRI at each post-operative follow-up. This outcome will assess, at a minimum, the following characteristics of the newly induced tissue: (i) presence or absence of a clear boundary between the device and the underlying tendon; (ii) presence or absence of a clear boundary between the newly induced tissue and the overlying deltoid muscle; (iii) maturation of newly induced tissue to resemble characteristics of underlying tendon tissue (versus debris or artifact).

# 4.3.3 Fill-In of Partial-Thickness Tears and Underlying Tendon Quality

For tendon defects treated by standalone use of the device (i.e., implantation without surgical repair using sutures/suture anchors), post-operative follow-up MRIs will be used to estimate the amount of defect fill-in with newly induced tissue and the quality of the filled-in tissue. In the absence of fill-in with newly induced tissue, defect progression (i.e., change in size relative to previous MRIs) will be assessed.

#### 4.3.4 Re-tear Rate

Re-tear following rotator cuff repair will be assessed at each follow-up visit using MRI. Any new observable defect (i.e. loss in supraspinatus tendon continuity) will be classified as a re-tear.

# 4.4 SECONDARY OUTCOME MEASURES

# **4.4.1** Safety

Safety will be evaluated by any of the following adverse events that occur over the duration of the study:

- 1. Any death
- 2. All serious adverse events (SAE) regardless of relation to the device or procedure
- 3. Any non-serious adverse event (AE) that is classified as either device or procedure-related
- 4. Any unanticipated adverse device effect (UADE)

Adverse events will be summarized by relation to the study devices or study procedure. Overall occurrence rate by event type will also be calculated.

# 4.4.2 Procedure Parameters

The following procedural parameters will be recorded on all subjects:

- 1. Device implant time: Mean ( $\pm$  SD) implant time defined as follows:
  - <u>Arthroscopic procedure</u>: Time from introduction of the guide wire instrument into the subacromial space to completion of last staple
  - <u>Mini-open procedure</u>: Time from introduction of the bioinductive implant into the subacromial space to completion of the last staple
- 2. Procedure technical success: The proportion of subjects where the device was successfully delivered and affixed to target tendon location.
- 3. Device implant position: An intra-operative photograph(s) or video recording showing the implant location of the device and all tendon and bone staples will be obtained.

# 4.4.3 Change in American Shoulder and Elbow Society (ASES) Scale

The mean ( $\pm$  SD) overall patient-reported ASES score (Range: 0 to 100) will be calculated at baseline and each subsequent follow-up. In addition, matched-pair analyses between baseline and successive follow-up visits will be performed to determine the mean ( $\pm$  SD) change in overall ASES score after surgery. Mean ( $\pm$  SD) overall shoulder pain from the ASES survey (Range: 0-10) will also be analyzed separately at baseline and each post-operative follow-up visit.

# 4.4.4 Change in Constant-Murley (Constant) Shoulder score

The mean ( $\pm$  SD) overall Constant score (Range: 0 to 100) will be calculated at baseline and each subsequent follow-up. In addition, matched-pair analyses between baseline and successive follow-up visits will be performed to determine the mean ( $\pm$  SD) change in overall Constant score after surgery. Mean ( $\pm$  SD) overall shoulder pain from the Constant survey (Range: 0-15) will also be analyzed separately at baseline and each post-operative follow-up visit.

# 4.4.5 Recovery

The following post-operative recovery parameters will be reported after discharge from the from study procedure:

- 1. Sling time: cumulative number of days (mean  $\pm$  SD) index shoulder is in a sling
- 2. Rehabilitation time: cumulative number of completed rehabilitation or physical therapy (PT) visits (mean  $\pm$  SD) to treat index shoulder
- 3. Return to work: cumulative number of days (mean  $\pm$  SD) between discharge and return to work (employed subjects only)
- 4. Return to normal daily activities (i.e. full, unrestricted activity): cumulative number of days (mean  $\pm$  SD) between discharge and return to normal daily activity

# 4.4.6 Subject Satisfaction

Subject satisfaction is a self-reported measure of satisfaction with the outcome of the index surgery. The level of satisfaction is assessed with a 5-point Likert scale. Each subject will also be asked to indicate whether (s)he would recommend the study procedure to a friend ("yes/no").

# 5 STATISTICAL ANALYSIS PLAN

# 5.1 Hypothesis Testing, Sample Size and Power

This is a single-arm, non-blinded study. The primary, quantitative endpoint is increase in thickness of the supraspinatus tendon at the device implant location.

The hypothesis being tested is that the overall thickness of the supraspinatus tendon increases by a minimum threshold identified as the objective performance criterion (OPC):

 $H_O$ :  $d \le OPC$  $H_A$ : d > OPC;

where "d" is the difference in supraspinatus tendon thickness at the location of the device at each follow-up interval (Follow-Up – Baseline).

Based upon finite element analysis (FEA) modelling, the theoretical reduction in tendon microstrains from the addition of 2 millimeters of new tendinous tissue at the tear site is 40% for articular-sided, partial thickness tears and 47% for bursal-sided tears. Data from clinical use of the device demonstrated a mean increase in tendon thickness of  $2.39 \pm 0.95$  millimeters at one year. <sup>13</sup>

Sample size was estimated using PASS 2008<sup>17</sup> and a one-sided one-sample t-test. The one-sided alpha level was set at 0.025. The value of d (mean of outcome measure) was set at 2 millimeters. Sample size calculations were made using powers of 80%, 85% and 90% and a one-sided alpha of 0.025 (non-inferiority; alpha-splitting) using a one-sample t-test.

Using a minimum OPC of 1.0 millimeter, a standard deviation of 1.0 millimeter, and 90% power, a total sample size of 13 subjects is adequate to test this hypothesis. Although adequate power is obtained with 13 subjects, to adjust for attrition and allow up to 30 evaluable subjects at 24-month follow-up meeting inclusion criterion 2A and another 30 evaluable subjects meeting inclusion criterion 2B, up to 150 subjects will be enrolled.

# 5.2 Interim Analyses

Interim analyses may be conducted any time to ensure site compliance with the protocol, evaluate outcomes, meet applicable reporting requirements (e.g., possible IRB annual reports, etc.), or present/publish interim results. Subgroup analyses may be performed to assess outcomes based upon subject demographics, type/size of rotator cuff tear, type of procedure performed, or other variables that may affect study outcomes. Additionally, analyses may be stratified by study site or Investigator as necessary to support Sponsor, Investigator, or site publication plans (Section 17).

# **6 ELIGIBILITY CRITERIA**

Subjects who meet all inclusion criteria (Section 6.1) and none of the exclusion criteria (Section 6.2) will be eligible to participate in the study.

Enrollment in the study occurs upon intra-operative confirmation that the subject meets all of the inclusion criteria and none of the exclusion criteria. Subjects who meet eligibility criteria and are enrolled will be followed per protocol through the end of the study (i.e., intent-to-treat). Subjects who do not meet the study eligibility criteria at the time of surgery will not be enrolled.

# 6.1 INCLUSION CRITERIA

Subjects enrolled in the study **MUST meet** all of the following criteria:

- 1. At least 21 years of age
- 2. Rotator cuff tear requiring surgery that meets either criterion A or B:
  - A. Medium or large partial-thickness tear or very small full-thickness tear of the supraspinatus tendon <u>planned for standalone treatment</u> (no surgical repair with sutures/suture anchors) <u>with the bioinductive implant</u>
  - B. Medium or large full-thickness tear primarily of the supraspinatus tendon <u>planned</u> for treatment with the bioinductive implant adjunctive to surgical repair
- 3. Chronic shoulder pain lasting longer than 3 months unresponsive to conservative therapy including, but not limited to, pain medication, physical therapy and injections
- 4. MRI of the shoulder within 60 days prior to the study procedure
- 5. Willing to comply with the prescribed post-operative rehabilitation program
- 6. Willing to be available for each protocol-required follow-up examination
- 7. Able to understand the informed consent process, including regulatory requirements such as HIPAA authorization, and document informed consent prior to completion of any study-related procedures
- 8. Ability to read, understand, and complete subject-reported outcomes in English

#### **6.2** EXCLUSION CRITERIA

Subjects enrolled in the study **MUST NOT meet** any of the following criteria:

- 1. Massive rotator cuff tears ( $\geq 5$  cm)
- 2. Acute rotator cuff tears less than 12 months from injury
- 3. Previous rotator cuff surgery on the index shoulder
- 4. Instability of the index shoulder
- 5. Chondromalacia of index shoulder ≥ Grade 3
- 6. Fatty infiltration of the index shoulder rotator cuff muscle  $\geq$  Grade 2

- 7. Calcification of the index shoulder rotator cuff
- 8. Genetic collagen disease
- 9. History of insulin dependent diabetes
- 10. History of auto-immune or immunodeficiency disorders
- 11. History of chronic inflammatory disorders
- 12. Oral steroid use in last 2 months or injectable steroid use in last 4 weeks
- 13. History of heavy smoking (> 1 pack per day) within last 6 months
- 14. Hypersensitivity to bovine-derived materials
- 15. Females of child-bearing potential who are pregnant or plan to become pregnant during the course of the study
- 16. Currently involved in any injury litigation or worker's compensation claims relating to the index shoulder
- 17. Enrolled, or plans to enroll, in another clinical trial during this study that would affect the outcomes of this study
- 18. History of non-compliance with medical treatment, physical therapy/rehabilitation, or clinical study participation
- 19. History of cognitive or mental health status that interferes with study participation

# 7 STUDY ASSESSEMENTS

The schedule of protocol-required study assessments is provided in **Table 7.1**. Adverse event (AE) reporting as required and defined in **Section 8** begins at the time of enrollment (i.e. intra-operative confirmation of eligibility) and concludes at the end of the study.

| | Baseline | Procedure | 3-Month | 1 Year | 2 Year |
|---|---|---|---|---|---|
| Study Evaluation | Within 60<br>Days of<br>Surgery | Within 60 Days of Baseline | ± 15 days | ± 45 days | ± 90 days |
| Informed Consent | <b>√</b> | | | | |
| Medical History & Exam | ✓ | | | | |
| Eligibility Assessment | ✓ | <b>√</b> 1 | | | |
| Enrollment (Date of Surgery) | | ✓ | | | |
| MRI | <b>√</b> <sup>2</sup> | | ✓2 | ✓2 | ✓2 |
| ASES Survey | <b>√</b> 3 | | <b>√</b> 3 | <b>√</b> 3 | <b>√</b> 3 |
| Constant-Murley Survey | ✓ | | ✓ | ✓ | ✓ |
| Procedure Data | | ✓ | | | |
| Medications | ✓4 | ✓4 | <b>√</b> 4 | <b>√</b> 4 | <b>√</b> 4 |
| Adverse Events | | <b>√</b> 5 | <b>√</b> 5 | <b>√</b> 5 | <b>√</b> 5 |
| Recovery/Satisfaction | | | ✓ | ✓ | ✓ |
| Questionnaire | | | | | |
| Revision/Additional | | | <b>√</b> 6 | <b>√</b> 6 | <b>√</b> 6 |
| Shoulder Surgery | | | | | |

**Table 7-1**: Schedule of Study Assessments

#### 7.1 ELIGIBILITY ASSESSMENT

Subjects are considered eligible for this study if they meet all of the inclusion criteria and none of the exclusion criteria as defined in **Section 6.1** and **Section 6.2**. The Investigator, co-Investigator, or sub-Investigator performing the study surgery will confirm eligibility at the time of the study surgery based upon intra-operative evaluation of the rotator cuff tear characteristics.

# 7.2 ENROLLMENT

Enrollment in the study occurs upon intra-operative confirmation that the subject meets all of the inclusion criteria and none of the exclusion criteria. Patients whose rotator cuff tears do not meet study eligibility criteria at the time of the study procedure will undergo tendon repair at the discretion of the surgeon (with or without use of the Rotation Medical Rotator Cuff System) and will not be enrolled in the study. Subjects who meet eligibility criteria will be considered enrolled into the study regardless of whether or not the device was successfully implanted. The date of the study surgery is

<sup>&</sup>lt;sup>1</sup>Eligibilty confirmation will be performed at the time of the study surgery to ensure the rotator cuff tear location/size meets eligibility criteria. Patients whose rotator cuff tears do not meet study eligibility criteria will not be enrolled in the study.

<sup>&</sup>lt;sup>2</sup>Each study MRI must be performed in accordance with the MRI study guideline.

<sup>&</sup>lt;sup>3</sup>The ASES-Patient Assessment is required. The ASES-Physician Assessment (ROM; strength) is optional as strength and ROM assessments are included in the Constant-Murley survey.

<sup>&</sup>lt;sup>4</sup>Only prescription medications to treat the index shoulder will be recorded.

<sup>&</sup>lt;sup>5</sup>Non-serious AEs will only be recorded if they are classified as either possibly or definitely related to either the study device or the study procedure.

<sup>&</sup>lt;sup>6</sup>Any additional surgical intervention performed on the index shoulder will be reported.

defined as the enrollment date and all subjects who are enrolled in the study will be followed per protocol unless voluntary consent is withdrawn. All subjects enrolled into the study will be identified through a unique identifier.

# 7.3 BASELINE ASSESSMENT

The following activities must be conducted within 60 calendar days prior to enrollment:

- 1. Obtain written informed consent.
- 2. Obtain a medical history.
- 3. Perform an MRI per the Sponsor imaging guidelines.
  - Provide the Sponsor with a de-identified digital copy of, or access to, the MRI.
- 4. Assess subject eligibility based on inclusion/exclusion criteria defined in **Section 6.1** and 6.2.
- 5. Administer the Constant-Murley shoulder survey.
  - Range of motion (ROM) should be measured with a goniometer and strength should be measured with a dynamometer.
- 6. Administer the ASES shoulder survey.
  - Completion of the ASES patient assessment section is required. Completion of the ASES physician assessment section is optional since ROM and strength are assessed during administration of the Constant-Murley survey.
- 7. Record prescription medications.
  - Record any prescription medications the subject is taking at the time of the baseline visit to treat his/her index shoulder.

All baseline assessments will be documented on their respective Case Report Forms (CRFs).

# 7.4 PROCEDURE ASSESSMENT

During the study procedure, use of any biological agents or implants aimed at augmenting tendon-to-bone healing, excluding the Rotation Medical Rotator Cuff System, are strictly prohibited. Intra-operative data along with the following study-specific procedure information will be documented on the Procedure CRF:

- 1. Device implant time
- 2. Procedure technical success
- 3. Device implant position
  - After implantation of the device, an intra-operative photograph(s) or video recording showing the implant location of the device and all tendon and bone staples will be obtained.
- 4. Intra-operative complication (if applicable; per Section 8)

Additionally, health insurance claim forms from the study surgical procedure (e.g., UB-04) will be collected by the Sponsor. Each claim form will be de-identified and serve as its own source document.

#### 7.5 PROCEDURE RULES

Subjects should be scheduled to undergo the study procedure within 60 days of baseline assessment. Device implantation will be performed in accordance with the Rotation Medical Rotator Cuff System device and instrument Instructions for Use (IFUs) and may

be performed as either a mini-open or arthroscopic procedure as determined by the surgeon and subject.

Subjects with medium or large partial-thickness tears or very small full-thickness tears of the supraspinatus tendon will undergo standalone device implantation without surgical repair of the tear.

Subjects with medium or large full-thickness tears primarily of the supraspinatus tendon will undergo device implantation adjunctive to surgical repair of the tear with sutures/suture anchors.

All subjects, regardless of supraspinatus tear size, will undergo acromioplasty and bursectomy. Removal of the periosteum at the lateral edge of the supraspinatus footprint is recommended to allow visualization of the footprint and facilitate proper device positioning. Debridement of the tendon may also be performed at the discretion of the surgeon.

Concomitant surgical treatment of the biceps tendon (i.e., tenotomy, tenodesis) and coracoacromial ligament (CA) release are also permitted during the study surgery at the discretion of the surgeon. If any other concurrent rotator cuff or shoulder surgeries not specified in this protocol are performed after the subject has been enrolled, a protocol deviation will be documented on the Protocol Deviation CRF. Wound closure is performed using standard methods.

If the physician determines intra-operatively that the rotator cuff tendon tear size or quality of tissue surrounding the tear does not meet study eligibility criteria, or determines additional concomitant surgery beyond what is permitted per protocol is required to provide the best surgical outcome for the subject, the subject will not be enrolled in the study.

#### 7.6 POST-OPERATIVE CARE

Post-operative care, including discharge instructions, pain management, and frequency/duration of physical therapy/rehabilitation regimen are at the discretion of the surgeon. To minimize the likelihood that the integrity or position of the device is compromised after implant, recommended rehabilitation guidelines are provided in **Table 7.2.** 

**Table 7-2**: Post-operative Rehabilitation Guidelines

| <b>Study Procedure</b> | Rehabilitation Guidelines |
|---|---|
| Device implant | Discard sling when comfortable |
| only; without | • Progression of motion as tolerated (Passive to Active Assisted to Active) |
| surgical repair | • 1st 4 Weeks: Forward flexion limited from 0° to 100° |
| | • 1st 6 Weeks: External rotation with arm by side (No ABER) |
| | • After 6 Weeks: No restrictions of motion or arm use |
| Device implant | Follow protocol for post-op surgical rotator cuff repair |
| with surgical | No additional requirements for the device |
| repair | • |

Subjects who undergo device implantation without rotator cuff repair should follow a rehabilitation course consistent with arthroscopic subacromial decompression (ASD) alone, but with limitations on forward flexion and external rotation in abduction (ABER). Subjects who undergo device implantation with cuff repair should follow a rehabilitation course consistent with standard rotator cuff repair.

# 7.7 FOLLOW-UP ASSESSMENTS

All subjects will undergo post-operative study assessments at 3 months, 1 year, and 2 years after discharge from the study procedure as described below and summarized in **Table 7.1**.

# 7.7.1 3-Month ( $\pm$ 15 Days) Follow-Up

- 1. Perform an MRI per the Sponsor imaging guidelines.
  - Provide the Sponsor with a de-identified digital copy of, or access to, the MRI.
- 2. Administer the Constant-Murley shoulder survey.
  - Range of motion (ROM) should be measured with a goniometer and strength should be measured with a dynamometer. NOTE: Strength or ROM testing at 3-Month Follow-Up may not be possible due to subject discomfort or ongoing rehabilitation and therefore missed or incomplete strength or ROM testing at this visit will not be considered as a protocol deviation.
- 3. Administer the ASES shoulder survey.
  - Completion of the ASES patient assessment section is required. Completion of the ASES physician assessment section is optional since ROM and strength are assessed during administration of the Constant-Murley survey.
- 4. Administer the recovery/satisfaction questionnaire.
- 5. Record prescription medications.
  - Record any prescription medications the subject is taking at the time of the follow-up visit to treat his/her index shoulder.
- 6. Record any new adverse events and update the status of any ongoing, previously-reported adverse events.
- 7. Report any new revision/additional shoulder surgeries performed on the index shoulder.

# 7.7.2 1-Year ( $\pm$ 45 Days) Follow-Up

- 1. Perform an MRI per the Sponsor imaging guidelines.
  - Provide the Sponsor with a de-identified digital copy of, or access to, the MRI.
- 2. Administer the Constant-Murley shoulder survey.
  - Range of motion (ROM) should be measured with a goniometer and strength should be measured with a dynamometer.
- 3. Administer the ASES shoulder survey.
  - Completion of the ASES patient assessment section is required. Completion of the ASES physician assessment section is optional since ROM and strength are assessed during administration of the Constant-Murley survey.
- 4. Administer the recovery/satisfaction questionnaire.
- 5. Record prescription medications.

- Record any prescription medications the subject is taking at the time of the follow-up visit to treat his/her index shoulder.
- 6. Record any new adverse events and update the status of any ongoing, previously-reported adverse events.
- 7. Report any new revision/additional shoulder surgeries performed on the index shoulder.

# 7.7.3 2-Year ( $\pm$ 90 Days) Follow-Up

- 1. Perform an MRI per the Sponsor imaging guidelines.
  - Provide the Sponsor with a de-identified digital copy of, or access to, the MRI.
- 2. Administer the Constant-Murley shoulder survey.
  - Range of motion (ROM) should be measured with a goniometer and strength should be measured with a dynamometer.
- 3. Administer the ASES shoulder survey.
  - Completion of the ASES patient assessment section is required. Completion of the ASES physician assessment section is optional since ROM and strength are assessed during administration of the Constant-Murley survey.
- 4. Administer the recovery/satisfaction questionnaire.
- 5. Record prescription medications.
  - Record any prescription medications the subject is taking at the time of the follow-up visit to treat his/her index shoulder.
- 6. Record any new adverse events and update the status of any ongoing, previously-reported adverse events.
- 7. Report any new revision/additional shoulder surgeries performed on the index shoulder.

The results of all follow-up assessments will be documented on their respective CRFs. Each reportable adverse event (**Section 4.1.1**) will be documented on an Adverse Event CRF.

# 7.8 UNSCHEDULED FOLLOW-UP

Any unscheduled return visits to the study center/Principal Investigator for non-standard of care evaluation for ongoing shoulder-related issues will be documented on a CRF. The reason for the visit and visit outcome will be documented. If an MRI, ASES survey, or Constant-Murley survey is completed, these assessments should also be documented on the appropriate CRFs. Visits required by the protocol or visits for routine post-operative follow-up are not considered unscheduled and do not need to be reported as an unscheduled visit.

# 7.9 REVISION/ADDITIONAL SHOULDER SURGERY

If the subject has additional or revision shoulder surgery on the index shoulder at any time during the follow-up period, the clinical site should make every effort to collect the procedure/operative notes for the procedure and complete the Revision/Additional Shoulder Surgery CRF. One (1) Revision/Additional Shoulder Surgery CRF should be completed for all surgeries performed on a single date. If a subject has multiple surgeries on the index shoulder on different dates, the Revision/Additional Shoulder Surgery CRF should be completed for each surgery date.

#### 7.10 EARLY WITHDRAWAL OR LOST TO FOLLOW-UP

If a subject wishes to withdraw from the study at any time, (s)he is able to do so voluntarily without having to justify it and without affecting her/his relationship with the Investigator.

Also, an Investigator may withdraw a subject from the study at any time if (s)he thinks it is in the subject's best interest.

The subject's future management will not be changed by a decision, voluntary or otherwise, to withdraw from the study.

All reasonable efforts should be made to retain the subject in this clinical study until completion of the clinical assessments at each follow-up visit. A subject will be considered "lost to follow-up" after a minimum of 2 documented phone calls to the subject were completed by a member of the study staff and a certified letter was sent to the last known address by a traceable method (e.g., certified mail; courier; commercial shipping/transport company).

Should subject early withdrawal or termination of participation occur, the termination information and the date of last contact with the subject should be recorded in the subject's records and included on the End of Study CRF.

# 7.11 END OF STUDY

Subjects will be exited upon successful completion of follow-up assessments or at the time of withdrawal or lost-to-follow-up. An End of Study CRF will be completed at the time of study completion or discontinuation.

# 8 ADVERSE EVENT DEFINITIONS AND REPORTING

Adverse events are to be reported from the time of enrollment through the last study follow-up visit.

# 8.1 DEFINITION OF ADVERSE EVENT (AE)

An Adverse Event (AE) is any undesirable clinical occurrence experienced by the subject. Any underlying disease that was present at the time of enrollment and prior to surgery (i.e. rotator cuff tendon tear) that persists after surgery is not considered an AE.

# 8.2 SERIOUS ADVERSE EVENT (SAE)

A Serious Adverse Event (SAE) includes any of the following events:

- Results in death
- Is life threatening
- Requires subject hospitalization or prolongation of existing hospitalization
- Requires invasive surgical intervention to fix the problem
- Results in persistent or significant disability/incapacity
- Is considered an important medical event

An important medical event that may not meet one of the above definitions might be considered as an SAE if it jeopardizes the health of the subject or requires surgical intervention to prevent one of the outcomes listed in the above definition. Elective hospitalization after the procedure that was planned prior to subject enrollment is not to be considered as an SAE.

# 8.3 UNANTICIPATED ADVERSE DEVICE EFFECT (UADE)

An Unanticipated Adverse Device Effects (UADE) is any serious adverse effect on health or safety, or any life-threatening problem or death caused by, or associated with, a device, if that effect was not previously identified in nature, severity, or degree of incidence in protocol, subject informed consent form, or application, or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects. Anticipated adverse events are listed as known risks in **Section 12.1**.

# 8.4 ASSESSING, RECORDING AND REPORTING AES, SAES, AND UADES

Only non-serious AEs that are classified by the Investigator as either device-related or procedure-related will be reported. All SAEs, regardless of relationship to the Rotation Medical Rotator Cuff System, and all UADEs will be reported.

An AE may be volunteered spontaneously by the subject or discovered as a result of questioning or physical examination by the Investigator or study staff. The following information should be reported on the Adverse Event CRF as soon as the Investigator becomes aware of the event and updated as needed until event resolves:

- Date of AE onset
- Date the Investigator became aware of the AE
- Main complaints/symptoms of the AE
- Relationship to the study device
- Relationship to the study procedure
- Status of the adverse event.

Source documents (e.g., procedural notes, treatment notes, or a signed clinical summary) may be required as supporting documentation for the reported AE.

# 9 MALFUNCTIONS

Failure of the Rotation Medical Rotator Cuff System to meet its performance specifications or to perform as intended will be documented on the Malfunction CRF. In the event of a malfunction, every effort must be made to return the suspected Rotation Medical device or instrument to the Sponsor for analysis. Malfunctions will be evaluated for reportable requirements through the FDA medical device reporting (MDR) system.

# 10 PROTOCOL DEVIATIONS

Investigators are required to adhere to the study protocol, signed Clinical Trial Agreement (CTA), applicable national or local laws and regulations, and any conditions required by the appropriate IRB/EC or applicable regulatory authorities.

A protocol deviation is used to describe situations in which the protocol was not followed (this includes all activities at each scheduled visit or activities occurring outside of the

study windows). All attempts should be made to obtain Sponsor approval of the deviation prior to their occurrence.

An Investigator must notify the Sponsor and the reviewing IRB/EC of any deviation from the Study Protocol that was done to protect the life or physical well-being of a subject (medical emergencies). Such notice should be given within 5 days of the occurrence. The Sponsor will determine if the subject affected is to continue in the study.

Documentation of deviations identified by the investigational center, the monitor, or other Sponsor representative(s) will be entered into the Protocol Deviation CRF for the purpose of tracking Investigator compliance with the protocol. The investigational center will be required to document actions taken to prevent recurrence of deviations. The Sponsor representative will initiate corrective actions based on individual deviations or trending reports as appropriate.

# 11 REPORTING REQUIREMENTS

**Table 11-1** shows a summary of all reporting requirements. In addition to this list, individual IRBs may add additional reporting requirements and/or require a different notification time frame.

**Table 11-1: Summary of Reporting Requirements** 

| Type of Report | Prepared by<br>Investigator FOR | Notification Time Frame |
|---|---|---|
| Death <sup>1</sup> | Sponsor & IRB | Within 24 hours of knowledge |
| Withdrawal of IRB approval | Sponsor | Within 5 working days of knowledge |
| Protocol Deviation to Protect<br>Subject Life or Physical<br>Well-Being | Sponsor & IRB | Within 5 working days of knowledge |
| Unanticipated Adverse<br>Device Effect (UADE) | Sponsor & IRB | Within 10 working days of knowledge |

<sup>&</sup>lt;sup>1</sup>Copies of death records, medical records for the events that led to the subject's death, a death certificate (if available), and an autopsy report (if performed) should be requested.

# 12 RISKS AND BENEFITS

#### 12.1 RISKS AND RISK MITIGATION

Study patients will be informed of all known potential side effects and complications associated with the study assessments and study procedure prior to enrollment in the study.

There are no known incremental risks to the subject for participating in the study. The risks associated with participating in this study are the same as if the patient is treated outside of the study using the same commercially-available device and include the following potential risks of rotator cuff surgery performed under general or regional anesthesia:

- Tissue inflammation
- The need for repeated surgery because tendons do not heal properly or tear again
- Pain or stiffness that won't go away
- Fever and/or infection
- Complication from anesthesia
- Nerve or blood vessel damage
- Adverse reaction to device

In addition, subjects will be required to undergo MR imaging. MRI is generally a well-tolerated procedure and there is no ionizing radiation involved with MR imaging. The potential risks are minimal and include claustrophobia, coil element heating and peripheral nerve stimulation, although the latter two are considered highly unlikely, given that the subjects will be imaged within preset safety guidelines to eliminate peripheral nerve stimulation. Coil element heating ranges from a mild sensation of heat to a potential burn. This is considered highly unlikely, as the coils have all undergone extensive testing and clinical use, and special pads are placed surrounding all contact points.

All Investigators will undergo training and subjects will be screened and evaluated for medical histories/conditions that may compromise safe, successful completion of any of the study assessments or performance of the device. Subjects with a known hypersensitivity to bovine-derived materials will not be enrolled in the study.

#### 12.2 BENEFITS

Participation in this study is voluntary. Subjects can obtain the same treatment without participating in this study. However, information gathered from this study will help the Sponsor to continue to evaluate long-term performance of the device when used alone or in conjunction with surgical repair to treat partial or full-thickness tears of the supraspinatus tendon.

# 13 DATA MANAGEMENT

# 13.1 DATA COLLECTION

Case report forms (CRFs) will be completed by the Investigator (or authorized study personnel) for each subject enrolled in the study. Data queries and edit checks will be used to reconcile discrepancies between data on the source documents and data entered on the CRFs. The Investigator must assure the accuracy and completeness of the recorded data. For the purpose of this study, the ASES and Constant shoulder surveys, as well as the Recovery/Satisfaction form, may act as their own source data.

# 13.2 DATA PROCESSING

All study documentation will be entered and maintained in a central database by the Sponsor or Sponsor-authorized representatives. Automatic and/or manual edit checks will be issued as necessary to correct discrepant data. Appropriate quality control measures will be established to ensure accurate and complete transfer of information from the study documentation to the central database. Data files will be exported from the central database for statistical analyses.

# 14 ADMINISTRATIVE RESPONSIBILITIES

The proposed study will be performed in accordance with all requirements set forth in the all applicable U.S. regulations, 21 Code of Federal Regulations (CFR) Parts 50 and 56, the World Medical Association Declaration of Helsinki, ISO 14155 (1) and (2), and any other applicable local laws and regulations.

#### 14.1 SITE AND INVESTIGATOR SELECTION

Each site and Investigator selected to participate will be evaluated to ensure each has the capacity, volume of surgical candidates, and capability to comply with all informed consent and protocol requirements. In addition, surgeon experience performing mini-open and arthroscopic surgeries to treat rotator cuff tears will be evaluated. Each study site and Investigator are required to comply with applicable local legal and regulatory requirements and applicable U.S. federal regulations.

# 14.2 TRAINING

All Investigators (Principal, co-Investigator, sub-Investigator) must be Board Certified orthopaedic surgeons with experience performing mini-open or arthroscopic rotator cuff repairs. Prior to first enrollment, each participating surgeon will complete Sponsor-provided training on the Rotation Medical Rotator Cuff System.

The Sponsor will also be responsible for ensuring each site and Investigator are properly trained on the study protocol and applicable regulatory requirements.

To insure uniform data collection and protocol compliance, the Sponsor or Sponsor-authorized representatives will train the Study Coordinator(s) and study staff on all components of the study including the study protocol, techniques for the identification of eligible subjects, instructions for data collection during the procedure, and schedules for follow-up.

# 14.3 INSTITUTIONAL REVIEW BOARD (IRB) / ETHICS COMMITTEE (EC)

It is the Investigator's responsibility to obtain and maintain written approval of the final study protocol and Informed Consent from the appropriate IRB or Ethics Committee. Investigators are responsible for submitting and obtaining initial and continuing review of the trial by their IRB/EC. It is also the Investigator's responsibility to notify the IRB/EC of any amendments to these documents. A copy of the written approval must be forwarded to the Sponsor prior to first device shipment. The written approval must identify the study and document the date of review.

The Investigators must keep on file all study-related correspondence with the IRB/EC and forward copies of such correspondence to the Sponsor.

# 14.4 INFORMED CONSENT FORM (ICF)

Informed consent must be obtained in accordance with the applicable guidelines on 21 CFR Part 50, current GCP, the Declaration of Helsinki, ISO 14155 (1) and (2), or local regulations and laws, whichever represents the greater protection of the individual. The subjects must be informed about their right to withdraw from the study at any time and for any reason without sanction, penalty, or loss of benefits to which the subject is otherwise entitled and also informed that withdrawal from the study will not jeopardize

their future medical care. The institutional standard subject consent form does not replace the study informed consent form (ICF).

The Sponsor will provide a study-specific template ICF to each site for IRB/EC submission. This template may be modified to suit the requirements of the individual study site. The Sponsor must pre-approve all changes to the ICF prior to initial submission to the IRB/EC. The Informed Consent Form must be approved by the IRB/EC prior to device shipment and a copy must be retained at the investigational site along with the other investigational forms. A signed copy of the consent form must be given to each subject enrolled in the study and a signed copy of the consent form must be retained for each subject at the investigational site.

Modifications to the study-specific Informed Consent Form and/or any written information distributed to subjects must be approved by the Sponsor, and the IRB/EC as necessary.

#### 14.5 CONFIDENTIALITY

All information and data sent to the Sponsor concerning subjects or their participation in this study will be considered confidential. All data used in the analysis and reporting of this evaluation will be used in a manner without identifiable reference to the subject. The Investigator consents to visits by the staff of the Sponsor and its authorized representatives and the U.S. FDA or any other local governmental body to review the study subjects' medical records, including any test or laboratory data that might have been recorded on diagnostic test media (e.g., MRI scan).

#### 14.6 AMENDING THE PROTOCOL

The Sponsor must write amendments in order to alter the protocol. Administrative changes that do not affect the subject benefit/risk ratio (e.g., editorial changes for clarity) may be implemented without any further approvals. Any change that would require alteration of the Informed Consent form must receive approval from all persons who approved the original protocol and from the IRB/EC prior to implementation. Following approval, the protocol amendment(s) will be distributed to all protocol recipients with instructions to append them to the protocol.

# 14.7 CRITERIA FOR TERMINATING STUDY

The Sponsor reserves the right to terminate the study early but intends only to exercise this right for valid scientific or administrative reasons or reasons related to the protection of study subjects. Investigators and associated IRB/EC will be notified in writing in the event of termination. Reasons for study termination include but are not limited to:

- The discovery of an unexpected, significant, or unacceptable risk to the study subjects.
- A decision on the part of the Sponsor to suspend or discontinue commercial distribution of the Rotation Medical Rotator Cuff System.

#### 14.8 CRITERIA FOR TERMINATING AN INVESTIGATIONAL CENTER

The Sponsor reserves the right to stop enrollment of subjects at an investigational center at any time for any of the following reasons including but not limited to:

• Repeated failure to complete case report forms (CRFs)

- Failure to obtain Informed Consent
- Failure to report any study subject deaths, SAEs, or UADEs within the timeframes specified in **Table 11-1**
- Repeated protocol deviations
- · Lack of study enrollment or study activity

#### 14.9 Sponsor Responsibilities

The Sponsor's responsibilities for this study are to:

- Provide sufficient training to support study activities per agreements executed with the study sites
- Select all clinical Investigators, study sites, and consultants (e.g., the study monitors) who participate in the study
- Provide financial support to each study site per agreements executed with the study sites
- Follow all regulatory standards per federal regulations for clinical study sites, core laboratories, and other participants, and ensure regular site monitoring to assure compliance with them
- Retain ownership of all clinical data generated in this study
- Work collaboratively with Investigators to present and publish study results

# 14.10 Investigator Responsibilities

The Investigator for each site is responsible for ensuring the study is conducted according to:

- All signed agreements
- The study protocol
- IRB/EC guidelines
- Applicable FDA regulations

The Investigator for each site may not begin enrollment until the Sponsor receives and approves (when necessary) required documents, including the complete signed Investigator Agreement, Protocol Signature Page, IRB/EC and ICF approvals.

It is acceptable for the Investigator to delegate one or more of the above functions to an associate or Co-Investigator or trained Study Coordinator; however, the Investigator remains responsible for the proper conduct of the clinical investigation, including obtaining the ICF, collecting all required data, submitting accurate and complete CRFs, etc.

At each site, appropriate procedures must be followed to maintain subject confidentiality according to HIPAA (Health Insurance Portability Accountability Assurance) regulations. Each site may have its own internal procedures or requirements for use and release of subject medical information in research studies. Each Investigator is responsible for obtaining appropriate approvals, consents or releases of medical information as dictated by their relevant subject privacy regulations.

The study is not transferable to other sites attended by the Investigator unless prior

approval is obtained from the appropriate IRB and the Sponsor.

# 15 MONITORING AND AUDITING

Monitoring visits to the investigational centers will be made frequently during the study to ensure that all aspects of the current approved protocol/amendment(s) are followed. Source documents will be reviewed for verification of agreement with data entered on the CRFs and all regulatory documents will be checked for accuracy including but not limited to IRB/EC approvals, study-related correspondence, and subject informed consent. The Investigator/institution guarantees direct access to source documents by designated Sponsor personnel and appropriate regulatory authorities. The site staff must agree to be available to meet with the Sponsor during each visit.

The study may also be subject to a quality assurance audit by the Sponsor or its designees as well as inspection by appropriate regulatory authorities.

# 16 REPORTS AND RECORDS

#### 16.1 REPORTS

Adverse events and Rotation Medical Rotator Cuff System malfunctions will be evaluated for reportable requirements through the FDA medical device reporting (MDR) system.

# 16.2 RECORDS

All records pertaining to the clinical study will be kept (in accordance with CFR §812.140 subpart d) for a minimum of 3 years following the date on which the study is terminated or completed.

If an Investigator wishes to withdraw from the responsibility of maintaining these study records, a transfer of that responsibility to a person willing to accept the responsibility (as outlined in CFR §812.140) must occur and be reported to the Sponsor not more than 10 days after the transfer occurs.

# 17 USE OF INFORMATION AND PUBLICATION

Any previously unpublished information provided to the Investigators by the Sponsor, such as patent applications, manufacturing processes and basic scientific data, is considered confidential and will remain the sole property of the Sponsor. The Investigator agrees to use this information only in accomplishing this study and will not use it for other purposes without the Sponsor's written consent.

An Investigator may publish the study experience from his/her site subject to approval by the Sponsor. The Sponsor will work collaboratively with Investigators to support data analyses for publication of study results. The Sponsor reserves the right to review all publications in order to verify accuracy of the data. The Investigator may proceed with the publication when notified by the Sponsor.

For any multi-center publications (if applicable), the number, names, and order of the authors will be determined by the Sponsor with input from the Investigators.

# 18 REFERENCES

1. Black EM, Higgins LD, Warner JJ. Value-based shoulder surgery: practicing outcomesdriven, cost-conscious care. J Shoulder Elbow Surg. 2013 Jul;22(7):1000-9.

- 2. Sher JS, Uribe JW, Posada A, Murphy BJ, Zlatkin MB. Abnormal findings on magnetic resonance images of asymptomatic shoulders. J Bone Joint Surg Am. 1995 Jan;77(1):10-5
- 3. Yamaguchi K, Ditsios K, Middleton WD, Hildebolt CF, Galatz LM, Teefey SA. The demographic and morphological features of rotator cuff disease. A comparison of asymptomatic and symptomatic shoulders. J Bone Joint Surg Am. 2006 Aug;88(8):1699-704.
- 4. Mall NA, Kim HM, Keener JD, Steger-May K, Teefey SA, Middleton WD, Stobbs G, Yamaguchi K. Symptomatic progression of asymptomatic rotator cuff tears: a prospective study of clinical and sonographic variables. J Bone Joint Surg Am. 2010 Nov 17;92(16):2623-33.
- 5. Kamath G, Galatz LM, Keener JD, Teefey S, Middleton W, Yamaguchi K. Tendon integrity and functional outcome after arthroscopic repair of high-grade partial-thickness supraspinatus tears. J Bone Joint Surg Am. 2009 May;91(5):1055-62
- 6. Kartus J, Kartus C, Rostgård-Christensen L, Sernert N, Read J, Perko M. Long-term clinical and ultrasound evaluation after arthroscopic acromioplasty in patients with partial rotator cuff tears. Arthroscopy. 2006 Jan;22(1):44-9.
- 7. Weber SC. Arthroscopic debridement and acromioplasty versus mini-open repair in the treatment of significant partial-thickness rotator cuff tears. Arthroscopy. 1999 Mar;15(2):126-31.
- 8. Bishop J, Klepps S, Lo IK, Bird J, Gladstone JN, Flatow EL. Cuff integrity after arthroscopic versus open rotator cuff repair: a prospective study. J Shoulder Elbow Surg. 2006 May-Jun;15(3):290-9.
- 9. Boileau P, Brassart N, Watkinson DJ, Carles M, Hatzidakis AM, Krishnan SG. Arthroscopic repair of full-thickness tears of the supraspinatus: does the tendon really heal? J Bone Joint Surg Am. 2005 Jun;87(6):1229-40.
- 10. Wolff AB, Sethi P, Sutton KM, Covey AS, Magit DP, Medvecky M. Partial-thickness rotator cuff tears. J Am Acad Orthop Surg. 2006 Dec;14(13):715-25.
- 11. Fuchs B, Gilbart MK, Hodler J, Gerber C. Clinical and structural results of open repair of an isolated one-tendon tear of the rotator cuff. J Bone Joint Surg Am. 2006 Feb;88(2):309-16.
- 12. Van Kampen C, Arnoczky S, Parks P, Hackett E, Ruehlman D, Turner A, Schlegel T. Tissue-engineered augmentation of a rotator cuff tendon using a reconstituted collagen scaffold: a histological evaluation in sheep. Muscles Ligaments Tendons J. 2013 Aug 11;3(3):229-35.
- 13. Data on file.
- 14. Richards RR, An KN, Bigliani LU, Friedman RJ, Gartsman GM, Gristina AG, Iannotti JP, Mow VC, Sidles JA, Zuckerman JD. A standardized method for the assessment of shoulder function. J Shoulder Elbow Surg. 1994 Nov;3(6):347-52.
- 15. Constant CR, Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res. 1987; 214: 160-64.
- 16. Chung SW, Park JS, Kim SH, Shin SH, Oh JH. Quality of life after arthroscopic rotator cuff repair: evaluation using SF-36 and an analysis of affecting clinical factors. Am J Sports Med. 2012 Mar;40(3):631-9.
- 17. Hintze, J. (2008). PASS 2008. NCSS, LLC. Kaysville, Utah, USA. www.ncss.com.